CLINICAL TRIAL: NCT01958008
Title: Randomized, Placebo-controlled, Double-blind Within Dose Groups, Multiple Rising-dose Study to Evaluate Safety, Tolerability, and PK of Oral BI 113608 Administered as Tablets Twice Daily Over 4 Weeks in Patients With COPD Associated With Chronic Bronchitis
Brief Title: BI 113608 Administered as Tablets Twice Daily Over 4 Weeks in Patients With Chronic Obstructive Pulmonary Disease Associated With Chronic Bronchitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 1314.5; 2012-005451-16 (EudraCT Number: EudraCT)
Record Dates: First submitted 2013-10-01; First posted 2013-10-08 (Estimated); Results first posted 2017-01-20 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2016-11

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

ARMS (3):
- BI 113608 low dose b.i.d. (Experimental): Film-coated tablet, oral administration with 240 mL water
  Interventions: Drug: Placebo to BI 113608 low dose b.i.d.; Drug: BI 113608 low dose b.i.d.
- BI 113608 medium dose b.i.d. (Experimental): Film-coated tablet, oral administration with 240 mL water
  Interventions: Drug: Placebo to BI 113608 medium dose b.i.d.; Drug: BI 113608 medium dose b.i.d.
- BI 113608 high dose b.i.d. (Experimental): Film-coated tablet, oral administration with 240 mL water
  Interventions: Drug: Placebo to BI 113608 high dose b.i.d.; Drug: BI 113608 high dose b.i.d.

INTERVENTIONS:
Drug: Placebo to BI 113608 high dose b.i.d. — Film-coated tablet
  Arms: BI 113608 high dose b.i.d.
Drug: Placebo to BI 113608 low dose b.i.d. — Film-coated tablet
  Arms: BI 113608 low dose b.i.d.
Drug: BI 113608 high dose b.i.d. — Film-coated tablet
  Arms: BI 113608 high dose b.i.d.
Drug: Placebo to BI 113608 medium dose b.i.d. — Film-coated tablet
  Arms: BI 113608 medium dose b.i.d.
Drug: BI 113608 low dose b.i.d. — Film-coated tablet
  Arms: BI 113608 low dose b.i.d.
Drug: BI 113608 medium dose b.i.d. — Film-coated tablet
  Arms: BI 113608 medium dose b.i.d.

SUMMARY:
The main objective of the current trial is to investigate safety, tolerability and pharmacokinetics of BI 113608 in COPD patients with symptoms of chronic bronchitis.

ELIGIBILITY:
Inclusion criteria:

1. All patients must sign an informed consent consistent with ICH-GCP guidelines and local legislations prior to any study-related procedures, which includes medication washout and restrictions.
2. All patients must have a documented diagnosis of COPD according to GOLD 2013.
3. Post-bronchodilator 50% = FEV1 < 80% of predicted at screening visit.
4. Post-bronchodilator FEV1/FVC <70% at screening visit.
5. Patients must have a history of chronic bronchitis as defined by symptoms of cough and sputum production on most days during at least three months for the past two consecutive years.
6. CAT Questionnaire at screening: a score of at least one for both cough (1st question) and sputum (2nd question).
7. Males and females between 40 and 80 years (inclusive) of age, on the day of patient´s signature of informed consent.
8. Patients must be current or ex-smokers with a smoking history of more than 10 pack years. Patients who have never smoked cigarettes must be excluded.
9. Patients must be able to perform technically acceptable pulmonary function tests (body plethysmography, forced spirometry and DLCO measurement).
10. Females must be of non-childbearing potential. Women of non-childbearing potential are defined as those who have undergone bilateral ovariectomy, bilateral salpingectomy or hysterectomy. If so, documentation confirming the surgical procedure must be available on the patient's source documents. A woman is also presumed to be infertile due to natural causes if she has been amenorrheic for more than 24 months. In questionable cases, a blood analysis of FSH and estradiol, which indicates the postmenopausal status according to the central laboratory ranges for postmenopausal females, is considered confirmatory.

Exclusion criteria:

1. Significant pulmonary disease other than COPD or other medical conditions* (as determined by medical history, examination, and clinical investigations at screening) that may, in the opinion of the investigator, result in the any of the following:

   1. Put the patient at risk because of participation in the study,
   2. Influence the results of the study,
   3. Cause concern regarding the patient's ability to participate in the study. (*e.g. cardiac, gastro-intestinal, hepatic, renal, metabolic, dermatologic, neurological, haematological, oncological and psychiatric; history of relevant orthostatic hypotension, fainting spells or blackouts; current chronic or relevant acute infections.)
2. Patients with any lung disease other than COPD (e.g. asthma, interstitial lung disease (ILD), cystic fibrosis, active tuberculosis, post-TB syndrome, clinically evident bronchiectasis, with a history of thoracotomy with pulmonary resection).
3. Patients with clinically relevant abnormal haematology, blood chemistry, or urinalysis at screening visit (Visit 1), if the abnormality defines a relevant disease as defined in exclusion criterion number 1.
4. All patients with a serum glutamate oxaloacetate transferase (SGOT) or serum glutamic pyruvic transaminase (SGPT) or total bilirubin higher than 1.5-fold ULN or serum creatinine higher than normal at Visit 1 (and at all repeated tests, if applicable) will be excluded regardless of the clinical condition. Laboratory evaluation can be repeated maximum two times.
5. A malignancy for which the patient has undergone resection, radiation therapy or chemotherapy within the last five years (patients with treated basal cell carcinoma are allowed).
6. Patients with current relevant psychiatric disorders based on the investigator´s judgement.
7. Patients with any respiratory infection (e.g. common cold, sinusitis, etc.) or COPD exacerbation within the six weeks prior to the screening visit (Visit 1) or between screening visit and randomization.
8. Patients with a history of two or more moderate or severe COPD exacerbations per year within the last two years.
9. Patients with a history of and/or active significant alcohol or drug abuse. See exclusion criterion number 1.
10. Patients who are being treated with non-permitted concomitant medication.
11. Patients with a recent history (i.e. three years or less) of heart failure or patients with any cardiac arrhythmia requiring drug therapy.
12. Patients who have previously been randomised in this trial.
13. Current participation in another clinical trial (as defined in the ICH Harmonised Tripartite Guideline for Good Clinical Practice (GCP)).
14. Donation of more than 100 mL of blood within the past four weeks prior to screening.
15. A history of additional risk factors for torsade-de-pointes (e.g., heart failure, relevant hypokalemia, family history of Long QT Syndrome).
16. Pregnant or nursing women.
17. Gastrointestinal tract surgery that might affect absorption and elimination of drugs.
18. Patients with known hypersensitivity / allergy to the investigational medicinal product (IMP) or its excipients.
19. Male Patients who do not agree to minimize the risk of female partners becoming pregnant from the first dosing day until two months after study completion.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2013-09; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (6):
- Germany (6):
  - Boehringer Ingelheim Investigational Site, Berlin
  - Boehringer Ingelheim Investigational Site, Frankfurt
  - Boehringer Ingelheim Investigational Site, Gauting
  - Boehringer Ingelheim Investigational Site, Großhansdorf
  - Boehringer Ingelheim Investigational Site, Lübeck
  - Boehringer Ingelheim Investigational Site, Mannheim

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial consisted of 3 sequential dose groups of 28 patients each. Within each dose group, 21 patients received BI 113608 and 7 received placebo
Groups:
- Placebo: Oral administration of Placebo matching BI 113608
- BI 113608 10 mg: Oral administration of BI 113608 10 mg film coated tablets twice daily
- BI 113608 25 mg: Oral administration of BI 113608 25 mg film coated tablets twice daily
- BI 113608 50 mg: Oral administration of BI 113608 50 mg film coated tablets twice daily
Period: Overall Study
Arm/Group | Placebo | BI 113608 10 mg | BI 113608 25 mg | BI 113608 50 mg
Started | 21 | 21 | 21 | 21
Completed | 20 | 21 | 20 | 21
Not Completed | 1 | 0 | 1 | 0
Not completed — Worsening of disease under study | 0 | 0 | 1 | 0
Not completed — Other adverse event | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set: All patients who received at least 1 dose of study drug were included in the Treated Set (TS).
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | BI 113608 10 mg | BI 113608 25 mg | BI 113608 50 mg | Total
Number analyzed (Participants) | 21 | 21 | 21 | 21 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.67 (6.64) | 58.90 (6.17) | 62.43 (7.21) | 60.38 (6.81) | 60.60 (6.71)
Gender [Count of Participants; unit: Participants]
  Female | 8 | 9 | 9 | 8 | 34
  Male | 13 | 12 | 12 | 13 | 50

OUTCOME MEASURES:

1. Primary Outcome: Number (%) of Patients With Drug-related Adverse Events (AEs)
Description: Number (%) of patients with drug-related adverse events (AEs)
Time Frame: AE's occuring upto end of treatment + 3 days follow up (Up to 31 days)
Population: Treated set (TS)
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | BI 113608 10 mg | BI 113608 25 mg | BI 113608 50 mg
Number analyzed (Participants) | 21 | 21 | 21 | 21
percentage of participants | 7 | 7 | 10 | 14

2. Secondary Outcome: Cmax,ss
Description: Cmax,ss (maximum measured concentration of BI 113608 in plasma at steady state over a uniform dosing interval tau)
Time Frame: Pre-dose and 0:15(hours:min),0:30,0:45,1:00,1:30,2:00,3:00,4:00,6:00,9:00,11:45,71:45,167:45,611:45,623:45,635:45,647:45,648:15,648:30,648:45,649:00,649:30,650:00,651:00,652:00,654:00,657:00,660:00,672:00,696:00,720:00 hours after drug administration
Population: Pharmacokinetic set (PKS): The patient set for the evaluation of PK endpoints included all evaluable patients in the treated set which provided at least 1 observation for at least 1 PK endpoint without important protocol violations relevant to the evaluation of PK.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | BI 113608 10 mg | BI 113608 25 mg | BI 113608 50 mg
Number analyzed (Participants) | 21 | 20 | 20
nmol/L | 44.1 (66.6) | 190 (45.1) | 328 (49.5)
Statistical Analysis 1: Comparison: BI 113608 10 mg vs BI 113608 25 mg vs BI 113608 50 mg; Dose proportionality was analysed over the dose range 10 to 50 mg for plasma PK parameters based on a power model; Test type: Superiority or Other; Regression, Linear; Power model that describes the functional relationship between the dose and pharmacokinetic endpoint Cmax,ss; Slope = 1.2674, 95% CI 2-sided [1.0636 to 1.4713], Standard Error of Mean 0.1019

3. Secondary Outcome: AUC Tau,ss
Description: AUC tau,ss (area under the concentration-time curve of the BI 113608 in plasma at steady state over a uniform dosing interval tau)
Time Frame: as for outcome 2
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | BI 113608 10 mg | BI 113608 25 mg | BI 113608 50 mg
Number analyzed (Participants) | 21 | 20 | 20
nmol*h/L | 166 (46.4) | 539 (43.3) | 1160 (42.3)
Statistical Analysis 1: Comparison: BI 113608 10 mg vs BI 113608 25 mg vs BI 113608 50 mg; Dose proportionality was analysed over the dose range 10 to 50 mg for plasma PK parameters based on a power model; Test type: Superiority or Other; Regression, Linear; Power model that describes the functional relationship between the dose and pharmacokinetic endpoint AUC tau,ss; Slope = 1.2139, 95% CI 2-sided [1.0519 to 1.3759], Standard Error of Mean 0.0810

4. Secondary Outcome: Tmax,ss
Description: Tmax,ss (time from last dosing to maximum concentration of the BI 113608 in plasma at steady state)
Time Frame: as for outcome 2
Population: PKS
Measure: Median (Full Range); unit: hours
Arm/Group | BI 113608 10 mg | BI 113608 25 mg | BI 113608 50 mg
Number analyzed (Participants) | 21 | 20 | 20
hours | 1.00 [0.50 to 2.03] | 0.750 [0.50 to 2.00] | 1.00 [0.50 to 3.00]

5. Secondary Outcome: T1/2,ss
Description: T1/2,ss (terminal half life of the BI 113608 in plasma at steady state)
Time Frame: as for outcome 2
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | BI 113608 10 mg | BI 113608 25 mg | BI 113608 50 mg
Number analyzed (Participants) | 21 | 20 | 20
hours | 17.4 (32.2) | 15.2 (14.9) | 16.2 (31.5)

6. Secondary Outcome: R(A,Cmax)
Description: R(A,Cmax) (accumulation ratio of the BI 113608 in plasma at steady state after multiple oral administration over a uniform dosing interval tau, expressed as ratio of Cmax at steady state and after first dose)
Time Frame: as for outcome 2
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | BI 113608 10 mg | BI 113608 25 mg | BI 113608 50 mg
Number analyzed (Participants) | 21 | 20 | 20
ratio | 1.36 (56.6) | 0.98 (42.2) | 1.13 (42.2)

7. Secondary Outcome: R(A,AUC)
Description: R(A,AUC) (accumulation ratio of the BI 113608 in plasma at steady state after multiple oral administration over a uniform dosing interval tau, expressed as ratio of AUC at steady state and after first dose)
Time Frame: as for outcome 2
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | BI 113608 10 mg | BI 113608 25 mg | BI 113608 50 mg
Number analyzed (Participants) | 21 | 20 | 20
ratio | 1.40 (35.8) | 1.20 (31.4) | 1.37 (27.0)

ADVERSE EVENTS:
Time Frame: From the first drug administration until 3 days after last study drug administration, up to 31 days.
Description: The above mentioned time frame corresponds to AEs that occurred during on treatment period
Groups:
- 10 mg Bid: Oral administration of BI 113608 10 mg film coated tablets twice daily
- 25 mg Bid: Oral administration of BI 113608 25 mg film coated tablets twice daily
- 50 mg Bid: Oral administration of BI 113608 50 mg film coated tablets twice daily
Arm/Group | Placebo | 10 mg Bid | 25 mg Bid | 50 mg Bid
Serious Adverse Events (participants affected / at risk) | 1/21 | 0/21 | 0/21 | 1/21
Other Adverse Events (participants affected / at risk) | 11/21 | 10/21 | 13/21 | 16/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=21) | 10 mg Bid (N=21) | 25 mg Bid (N=21) | 50 mg Bid (N=21)
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 0
Blood potassium increased (Investigations) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=21) | 10 mg Bid (N=21) | 25 mg Bid (N=21) | 50 mg Bid (N=21)
Nasopharyngitis (Infections and infestations) | 1 | 2 | 2 | 3
Conjunctivitis (Infections and infestations) | 2 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 2 | 2 | 2 | 0
Headache (Nervous system disorders) | 2 | 4 | 4 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 1 | 3
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 3
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 3 | 3 | 5
Nausea (Gastrointestinal disorders) | 0 | 3 | 2 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 1 | 2 | 0
Vomiting (Gastrointestinal disorders) | 1 | 2 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.